CLINICAL TRIAL: NCT07123883
Title: Dry Needle Treatment for Acute Temporomandibular Disorders (TMD): A Clinical Perspective
Brief Title: Dry Needling for Temporomandibular Disorder
Acronym: DN-TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Atlas E-22686390-050.99-72665; Atlas E-22686390-050.99-72665 (Other Grant/Funding Number: Atlas University)
Record Dates: First submitted 2025-07-21; First posted 2025-08-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: TMD/Orofacial Pain; Muscle Spasm
Keywords: Dry needling; Temporomandibular Disorders; Muscle Pain Dysfunction
MeSH Terms: conditions — Spasm; Temporomandibular Joint Disorders | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: All participants in the study were randomly assigned to one of two groups: the dry needling group (DNG) or the sham needling group (SG). In the DNG, deep dry needling was administered to the most sensitive myofascial trigger point identified in either the masseter or anterior temporalis muscle using a sterile acupuncture needle (0.20 × 13 mm, Qinzhou, China). The procedure was performed by a physiotherapist with seven years of clinical experience, under the supervision of a licensed physician.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling Group (DNG) (Experimental): In the DNG, under aseptic conditions, the needle was inserted into the predetermined trigger point of the masseter muscle using a guide tube. It was then advanced deeply into the muscle tissue and manipulated using a pistoning technique involving approximately ten in-and-out movements without complete withdrawal. The direction of the needle was systematically varied to stimulate adjacent regions of the muscle, maintaining an average insertion rate of one movement per second. Local twitch responses (LTRs) were elicited and monitored throughout the procedure. Upon completion, the needle was withdrawn, and gentle pressure was applied to the insertion site with a sterile cotton pad to prevent bleeding
  Interventions: Procedure: Dry Needling
- Sham Group (SG) (Sham Comparator): In the SG, a validated sham needling procedure was simulated. Participants were positioned identically to the DNG and the same type of needle and guide tube were used. However, the safety lock on the needle was left intact, preventing skin penetration. A cotton pad was applied with light pressure to the skin surface, mimicking the procedure used in the DNG. This approach has been previously validated as a reliable sham control in dry needling research
  Interventions: Other: sham needling

INTERVENTIONS:
Procedure: Dry Needling — Dry Needling
  Arms: Dry Needling Group (DNG)
Other: sham needling — In the SG, a validated sham needling procedure was simulated.
  Arms: Sham Group (SG)

SUMMARY:
This randomized controlled trial investigates the clinical effectiveness of dry needling in individuals with myofascial temporomandibular disorder (TMD). The study compares dry needling applied to trigger points in the masseter and temporalis muscles with conventional physical therapy. Primary outcomes include changes in pain intensity, and muscle EMG. Given these considerations, this study aims to investigate the clinical acute effectiveness of dry needling applied to the masseter and temporalis muscles in individuals diagnosed with myofascial TMD.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMDs) are a common group of musculoskeletal conditions affecting the jaw joint and surrounding muscles, often characterized by pain, limited mandibular mobility, and muscle tenderness. Among the various subtypes of TMD, myofascial pain is the most prevalent and typically involves the presence of myofascial trigger points (MTrPs) in the masticatory muscles. Dry needling (DN) is a minimally invasive technique that targets MTrPs using monofilament needles to induce a local twitch response and disrupt dysfunctional motor end plate activity.

This single-blinded, randomized controlled trial aims to evaluate the acute clinical effectiveness of DN compared to conventional physical therapy in individuals with myofascial TMD. In our study, 36 participants were randomly assigned to one of two groups: the dry needling group or the sham group, using a randomization process conducted through random.org. The study aimed to examine the acute effects following a single application. A double-blind design was employed, with separate physiotherapists responsible for administering the intervention and conducting the assessments. The study consisted of three stages: pre-intervention assessment, intervention, and post-intervention assessment.

Jaw pain intensity was evaluated at the end of the range of motion using a 100 mm VAS, a tool recognized for its high reliability in musculoskeletal assessments. All participants were asked to indicate their pain level on the VAS, allowing for a subjective quantification of perceived pain intensity

Surface electromyographic (sEMG) activity of the jaw muscles was recorded bilaterally from the anterior temporalis (TA-R, TA-L) and masseter (MM-R, MM-L) muscles using the BioPAK System (version 7.2; BioResearch Associates Inc., Milwaukee, WI, USA).

ELIGIBILITY:
Inclusion Criteria

* Patients aged between 18 and 45 years presenting with complaints of jaw pain to the Department of Dentistry at A University.
* Diagnosed with myofascial pain associated with temporomandibular dysfunction by a dentist, based on the Axis I criteria of the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD).
* Jaw pain persisting for at least three months.
* Pain elicited upon palpation of the masseter and/or temporalis muscles.
* Presence of clicking or crepitus in the temporomandibular joint during mandibular movements.
* Self-reported jaw muscle fatigue or stiffness, particularly upon awakening. Exclusion Criteria
* History of any confirmed or suspected inflammatory or neurological condition.
* Presence of any oral or dental infection.
* Any cognitive or communication impairment affecting data collection.
* History of head or facial trauma.
* Allergy to metals.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-05-18 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Jaw pain intensity | Baseline and After 10-minute
  Jaw pain intensity was evaluated at the end of the range of motion using a 100 mm VAS, a tool recognized for its high reliability in musculoskeletal assessments. All participants were asked to indicate their pain level on the VAS, allowing for a subjective quantification of perceived pain intensity . Pain intensity was assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain), with higher scores indicating worse outcomes.

SECONDARY OUTCOMES:
Surface electromyographic (sEMG) | Baseline and After 10-minute
  Surface electromyographic (sEMG) activity of the jaw muscles was recorded bilaterally from the anterior temporalis (TA-R, TA-L) and masseter (MM-R, MM-L) muscles using the BioPAK System (version 7.2; BioResearch Associates Inc., Milwaukee, WI, USA).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Faculty of Dentistry, Atlas University, Istanbul, Istanbul
  - Istanbul Atlas University, Faculty of Dentistry, Istanbul, Kagithane

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared due to privacy and confidentiality concerns and because data sharing is not required for the objectives of this study.